CLINICAL TRIAL: NCT06878703
Title: Efficacy of Dexmedetomidine Versus Midazolam Sedation on Extubation Time in Mechanically Ventilated Preterm Infants: a Randomized Controlled Multicenter Trial - DEXPRE
Brief Title: Efficacy of Dexmedetomidine Versus Midazolam Sedation on Extubation Time in Mechanically Ventilated Preterm Infants
Acronym: DEXPRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: DrData (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: APHP230813
Record Dates: First submitted 2025-02-21; First posted 2025-03-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: PreTerm Neonate; Sedation for Invasive Mechanical Ventilation; Very Preterm Neonates With Sedation for Invasive Mechanical Ventilation
Keywords: Mechanical ventilation; Sedative agent; Sedation-analgesia; Midazolam; Extubation; Very preterm neonate; Dexmedetomidine
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam (Active Comparator): In the control group, neonates will receive midazolam intravenously, starting with a 10 μg/kg loading dose over 30 minutes, followed by a maintenance dose of 10-40 μg/kg/h.
  Interventions: Drug: Midazolam
- Dexmedetomidine (Experimental): In the experimental group, neonates will receive continuous intravenous administration of dexmedetomidine, with a loading dose of 0.05 μg/kg over 30 minutes followed by a continuous maintenance dose (from 0.05 to 0.2 μg/kg/hour).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — Continuous intravenous administration with a loading dose of 10 µg/kg over 30 min, followed by a maintenance dose (from 10 to 40 µg/kg/h)
  Arms: Midazolam
Drug: Dexmedetomidine — Continuous intravenous administration with a loading dose of 0.05 μg/kg over 30 minutes followed by a maintenance dose (from 0.05 to 0.2 μg/kg/h)
  Arms: Dexmedetomidine

SUMMARY:
Very preterm neonates (born before 32 weeks' gestation) often require invasive mechanical ventilation (IMV) to manage respiratory insufficiency. In France, around 8,250 infants are born annually at <32 weeks, with an estimated 5,000 needing IMV. Although non-invasive support such as continuous positive airway pressure (CPAP) has become more common, a substantial proportion of these neonates still transition to IMV within the first few days of life. To reduce lung injury and the incidence of bronchopulmonary dysplasia (BPD), a key strategy in neonatal intensive care involves limiting the duration of IMV and promoting earlier extubation.

However, effective sedation and analgesia are essential for preterm infants subjected to intubation and mechanical ventilation. Traditionally, neonatologists combine a sedative (frequently midazolam) with an opioid (morphine, fentanyl, or sufentanil). Although these agents control pain and distress, they may cause respiratory depression, complicate weaning, and potentially contribute to adverse long-term outcomes. Midazolam, one of the few sedatives authorized for use in neonates, can improve comfort and sedation scores, but concerns persist about hypotension, altered cerebral perfusion, and a possible link to intraventricular hemorrhage (IVH). Moreover, combining benzodiazepines and opioids can prolong ventilation, increase the risk of complications, and impede timely extubation.

Rationale for Dexmedetomidine (DEX) Dexmedetomidine (DEX) is a highly selective α2-adrenergic agonist that offers sedative, anxiolytic, and analgesic properties with relatively minimal respiratory depression. Unlike certain other sedatives, DEX induces a state akin to natural sleep, allowing for easier arousal and potentially better respiratory drive. Animal studies suggest that DEX might be neuroprotective, reducing inflammation, oxidative stress, and apoptotic processes that can be detrimental to the developing brain. These features make DEX a promising alternative to the commonly used benzodiazepine-opioid regimens in very preterm neonates, who remain especially vulnerable to adverse drug effects.

Minimizing Invasive Mechanical Ventilation Reducing the time on IMV is crucial for preventing ventilator-induced lung injury and decreasing the likelihood of BPD. Early extubation is a central goal in this population, but sedation-related respiratory depression can thwart successful weaning and lead to reintubation. By preserving spontaneous breathing more effectively than midazolam or high-dose opioids, DEX may help neonates maintain adequate ventilation as they transition to non-invasive support. Furthermore, DEX's analgesic action could reduce the need for opioids, thereby mitigating withdrawal risks and other opioid-related complications such as feeding intolerance and extended hospital stays.

Objective of the DEXPRE Trial The objective of the DEXPRE trial is to compare the efficacy of dexmedetomidine-based sedation with that of midazolam-based sedation in very preterm neonates requiring IMV. Specifically, investigators aim to determine whether DEX can facilitate more rapid extubation and better overall respiratory outcomes compared to midazolam. By systematically evaluating sedation quality, respiratory stability, and potential side effects, the trial seeks to generate evidence that will guide future sedation protocols in neonatal intensive care units.

DETAILED DESCRIPTION:
Hypothesis : the use of dexmedetomidine (DEX), 0.05 to 0.2 μg/kg/h, for very preterm neonates (<32 weeks' gestation, WG), requiring prolonged sedation throughout the period of invasive mechanical ventilation (IMV) (usually after intubation and until extubation), may improve weaning, and thus reduce extubation time in neonatal intensive care units.

Population of study participants : Very preterm neonate (gestational age at birth < 32 WG) with corrected gestational age <45 WG).

In the experimental group, neonates will receive dexmedetomidine via continuous intravenous infusion, starting with a 0.05 μg/kg loading dose over 30 minutes, followed by a maintenance dose ranging from 0.05 to 0.2 μg/kg per hour.

In the control group, neonates will receive midazolam via continuous intravenous infusion, starting with a 10 μg/kg loading dose over 30 minutes, followed by a maintenance dose ranging from 10 to 40 μg/kg per hour.

To achieve the randomization of 292 patients, an estimated enrollment of about 380 participants is anticipated, resulting in an allocation of 146 patients per study arm.

During the inclusion visit, after verifying the inclusion and exclusion criteria, an investigator will inform the parents of eligible neonates. If the neonate requires invasive mechanical ventilation and meets the randomization criteria, the investigator will proceed with the randomization.

According to the allocation arm, the nurse in charge of the patient will be able to prepare the experimental treatment using the kit provided by the hospital pharmacy.

The experimental treatment will start with a 30-minute loading dose, followed by a maintenance dose. The infusion rate will be adjusted according to medical prescriptions to achieve the desired sedation level, ranging from 0.1 mL/hr to 0.4 mL/hr. This treatment can be administered via any venous line, either peripheral or central.

Vital signs will be regularly recorded at 5, 10, 30, and 60 minutes, then at 2, 3, 6, and 12 hours after the start of treatment. Following this, recordings will be taken every 12 hours until the treatment ends.

Pain scores will be recorded 30 and 60 minutes after the initiation of treatment, and then every 3 hours, following standard practice.

On the day of extubation, routine data recording will include the timing and duration of experimental treatment and opioid interruptions, the extubation time, vital signs before and after treatment discontinuation, and any adverse events.

The final study visit will occur when the child reaches 2 years of corrected age +/- 2 months. At this visit, weight, height, head circumference, cerebral palsy status, age of walking acquisition, and the Ages & Stages Questionnaire (ASQ) score will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in NICU (intubated or not yet),
* Gestational age at birth < 32 weeks of gestation (WG),
* Corrected gestational age <45 weeks postmenstrual age Written or electronic informed consent signed by both parents.

Randomization Criteria :

* Indication for sedation in the context of invasive mechanical ventilation,
* Patient intubated or not yet,
* Elective sedation (acceptable delay between the decision to sedate and the administration of the sedative agent),
* Presence or plan of a venous access,
* No medical contraindication related to the administration of dexmedetomidine or midazolam,
* No previous use of dexmedetomidine or midazolam within 48 hours, except for the sedation procedure for intubation,
* No concomitant use of curare agent,
* No clonidine treatment,
* No previous extubation within 7 days,
* No hemodynamic instability
* No palliative care,

Exclusion Criteria:

* Patient admitted in NICU (intubated or not yet),
* Gestational age at birth < 32 weeks of gestation (WG),
* Corrected gestational age <45 weeks postmenstrual age Written or electronic informed consent signed by both parents.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-10-16 (Estimated)

PRIMARY OUTCOMES:
Time, measured in minutes, is evaluated from the discontinuation of the experimental treatment (either dexmedetomidine-based or midazolam-based sedation) to extubation. | from the discontinuation of the experimental treatment to extubation (48 maximum)
  to compare the efficacy of dexmedetomidine-based sedation versus midazolam-based sedation in very preterm neonates.

SECONDARY OUTCOMES:
Administration of Opioid Agents During Sedation with Dexmedetomidine or Midazolam in Neonatal Intensive Care. | from the start of treatment (dexmedetomidine or midazolam) until extubation (16 days maximum)
  Administration of opioid agents during the period of interest, i.e., from the start of treatment (DEX or midazolam) until extubation (total cumulative dose and morphine equivalents in mg/kg, duration). opioids include morphine (1), fentanyl (0.010), remifentanil (0.15), sufentanil (0.003) and methadone (0.3).
Quality of sedation | Before sedation, then every 30 min after sedation initiation, then every 3 hours after the initial 60 min, and up to 14 days
  Time (in hours) between start of sedation and achievement of a normal Comfort B score (ie. between 11 and 17),
Extubation failure 24 hours after extubation | In 24 hours after extubation
  Intubation proportion at 24 hours after extubation.
Withdrawal syndrome (Finnegan score >8). | 6 hours, within 7 days after extubation.
  Proportion of patients with at least one value of the Finnegan score > 8 from within 3 days after extubation.
Hemodynamic and respiratory adverse effects between inclusion and 84 hours after treatment discontinuation, | From start of the sedation until 84 h after the sedative is stopped (maximum 18 days)
  * Bradycardia defined by heart rate < 80 bpm considered as clinically significant by the treating physician, despite optimization of hemodynamic management
  * Hemodynamic instability defined by a mean blood pressure below corrected GA, or a skin recoloration time > 3 seconds despite optimization of haemodynamic management
  * Desaturation <85% despite optimization of mechanical ventilation
  * Reintubation
In hospital morbi mortality. | the period of hospitalization and within the limit of 24 months
  Severe neonatal morbidity as :
  * late onset sepsis defined by a positive blood culture and antibiotic therapy more than 72 hours,
  * necrotizing enterocolitis according to Bell's definition61
  * moderate (fraction of inspired oxygen (FiO2) <30%) and severe (FiO2 ≥30%) bronchopulmonary dysplasia at 36 WG defined by need of IMV, nasal continuous positive airway pressure, or nasal cannula at 36 weeks postmenstrual age, according to Jobe's definition
  * retinopathy of prematurity is diagnosed at the fundus performed systematically before discharge, intraventricular hemorrhage diagnosed on routine transfontanelar ultrasound, according to Papile classification

OTHER OUTCOMES:
Exploratory outcome: Duration (in hours) of invasive mechanical ventilation from intubation to extubation | From intubation to extubation
  To assess the impact of the treatment on Duration of mechanical ventilation
Exploratory outcome: Length of stay in the NICU | Within the limit of 24 months
Exploratory outcome: : Short-term clinical outcomes | at 36 Week of Gestation
  Survival without moderate and severe bronchopulmonary dysplasia at 36 WG,
Exploratory outcome: 2 years neurodevelopment | At 2 years
  Neurodevelopment at 2 years assessed by the Score of Ages & Stages (ASQ) at 2 years.
  Score of Age and Stages (ASQ)
  Questionnaire composed of five fields (communication, gross motor skills, fine motor skills, problem solving and individuals or social skills) ; for each field :
  Minimum value is 0 Maximum value is 60 An Higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Clément CHOLLAT, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Armand Trousseau, APHP Service : Department of Neonatology, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided